CLINICAL TRIAL: NCT00006006
Title: Thalidomide for Unresectable Hepatocellular Cancer With Optional Interferon Alpha-2a Upon Disease Progression
Brief Title: Thalidomide Plus Interferon Alfa in Treating Patients With Progressive Liver Cancer That Cannot be Surgically Removed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02347; NYU-9938; NCI-101; CDR0000068014 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2003-09

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Interferon-alpha; Thalidomide

ARMS (1):
- Arm I (Experimental): Patients receive oral thalidomide once daily. Patients on a stable dose of thalidomide for at least 4 weeks with evidence of progressive disease receive interferon alfa subcutaneously twice daily. Treatment continues in the absence of disease progression after initiation of interferon alfa therapy or unacceptable toxicity.
  Interventions: Biological: recombinant interferon alfa; Drug: thalidomide

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: thalidomide

SUMMARY:
Phase II trial to study the effectiveness of thalidomide plus interferon alfa in treating patients who have progressive liver cancer that cannot be surgically removed. Thalidomide may stop the growth of liver cancer by stopping blood flow to the tumor. Interferon alfa may interfere with the growth of the cancer cells. Combining thalidomide and interferon alfa may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the feasibility and activity of thalidomide in patients with unresectable hepatocellular carcinoma.

II. Evaluate the toxicity of thalidomide in these patients. III. Assess the use of interferon alfa in patients who develop disease progression while being treated with thalidomide.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily. Patients on a stable dose of thalidomide for at least 4 weeks with evidence of progressive disease receive interferon alfa subcutaneously twice daily. Treatment continues in the absence of disease progression after initiation of interferon alfa therapy or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatocellular carcinoma OR
* Diagnosis of hepatocellular carcinoma based on characteristic mass and alpha-fetoprotein greater than 500 in the setting of known cirrhosis or chronic hepatitis B or C
* Measurable disease

  * At least 20 mm in one dimension
* Not amenable to curative surgical resection

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Hematopoietic:

* Absolute neutrophil count greater than 1,200/mm^3
* Hemoglobin at least 8.0 mg/dL
* Platelet count at least 25,000/mm^3

Hepatic:

* Bilirubin no greater than 5 mg/dL
* Liver function tests no greater than 5 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Regardless of fertility status:

  * All women (unless they have undergone hysterectomy or have been amenorrheic or postmenopausal for at least 2 years) must use at least 1 highly active method of contraception AND 1 additional effective method of contraception at least 4 weeks before, during, and for at least 4 weeks after study
  * All men (even if they have undergone a successful vasectomy) must use effective barrier contraception during and for at least 4 weeks after study
* No other medical condition that would preclude study
* No other prior malignancy in past 5 years except curatively resected basal cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior biologic therapy regimen
* No prior interferon or thalidomide for hepatocellular cancer

Chemotherapy:

* No more than 1 prior chemotherapy regimen

Other:

* No concurrent barbiturates or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2000-08; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D. Volm, MD, Study Chair — NYU Langone Health
Locations (2):
- United States (2):
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York

REFERENCES:
- [Result] Schwartz JD, Sung M, Schwartz M, Lehrer D, Mandeli J, Liebes L, Goldenberg A, Volm M. Thalidomide in advanced hepatocellular carcinoma with optional low-dose interferon-alpha2a upon progression. Oncologist. 2005 Oct;10(9):718-27. doi: 10.1634/theoncologist.10-9-718. PMID 16249352